CLINICAL TRIAL: NCT03175978
Title: Pilot Study of IGF-Methotrexate Conjugate in the Treatment of Myelodysplastic Syndrome, CMML and Oligoblastic AML
Brief Title: IGF-MTX Conjugate in the Treatment of Myelodysplastic Syndrome
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Funding
Sponsor: IGF Oncology, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AML-03
Record Dates: First submitted 2017-05-25; First posted 2017-06-05 (Actual); Results first posted 2024-05-21 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Chronic; Anemia, Refractory, With Excess of Blasts
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Chronic; Anemia, Refractory, with Excess of Blasts

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- IGF/MTX (Experimental): This arm will evaluate use of IGF-Methotrexate conjugate (765IGF-MTX) in patients with advanced, previously treated MDS, CMML and O-AML. 765IGF-MTX at a dose of 0.20 to 2.5 µequivalents per kg is administered as an IV infusion over 1.5 hours on days 1, 8 and 15 of a 28 day cycle. Treatment continues until disease progression, as assessed after 2 cycles, unacceptable toxicity, or patient refusal.
  Interventions: Drug: IGF/MTX

INTERVENTIONS:
Drug: IGF/MTX — 765IGF-MTX is supplied as a 5 ml sterile solution at 4.0 µeq per ml 765IGF-MTX concentration in aqueous 10 mM HCl in a 10 ml glass vial
  Other Names: insulin-like growth factor-1/methotrexate conjugate; 765IGF-methotrexate

SUMMARY:
The primary objective of this study is to determine the safety and tolerability of utilizing the insulin-like growth factor-1-methotrexate conjugate, 765IGF-MTX for the treatment of advanced, previously treated myelodysplastic syndrome (MDS), chronic myelomonocytic leukemia (CMML) and oligoblastic acute myelogenous leukemia (oligoblastic AML or O-AML), including determining the maximum tolerated dose (MTD).

DETAILED DESCRIPTION:
This pilot study will evaluate use of IGF-Methotrexate conjugate (765IGF-MTX) in patients with advanced, previously treated MDS, CMML and O-AML. 765IGF-MTX at a dose of 0.20 to 2.5 µequivalents per kg is administered as an IV infusion over 1.5 hours on days 1, 8 and 15 of a 28 day cycle. Treatment continues until disease progression, as assessed after 2 cycles, unacceptable toxicity, or patient refusal. Assessment of response will be confirmed by bone marrow studies performed at the end of cycles 2, 4, and 6 (each +/- 3 days).

Pharmacokinetics will be performed before and for up to 24 hours after drug administration on days 1 (for 24 hrs) and 15 (for 24 hrs) of cycle 1. Pharmacodynamic samples will be assessed pre-dosing on day 1 of cycle 1, pre-dosing on days 1 and 15 of cycle 2, and pre-dosing on day 15 of cycles 4 and 6.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of O-AML that is refractory to or intolerant to standard therapy and is no longer likely to respond to such therapy (at least one line of therapy); or Diagnosis of MDS/CMML that is refractory to or intolerant to standard therapy and is no longer likely to respond to such therapy (at least one line of therapy)
* Confirmed histologic diagnosis on bone marrow biopsy and aspirate within 28 days of trial entry prior to starting cycle 1.
* Platelets > 10 x 10^9/L
* ECOG performance status of 0, 1 or 2
* Prior systemic chemotherapy, immunotherapy, or biological therapy, radiation therapy and/or surgery are allowed; prior use of systemic methotrexate > 1 month prior to study entry is allowed. Intrathecal methotrexate is allowed prior to and during treatment per investigator discretion.
* Patient must have recovered from the acute toxic effects (≤ grade 1 CTCAE v.4.0) of previous anti-cancer treatment prior to study enrollment; the only exception is that grade 2 neuropathy is permitted
* Adequate organ function within 14 days of study registration
* Negative serum pregnancy test in females. Male and female patients with reproductive potential must use an approved contraceptive method if appropriate

Exclusion Criteria:

* ECOG PS >2.
* Patients with active extramedullary disease.
* Pleural effusions or ascites.

  * Grade 3 peripheral neuropathy within 14 days before enrollment.
* Active uncontrolled infection or severe systemic infection (enrollment is possible after control of infection).
* Myocardial infarction within ONE months prior to enrollment or has New York Heart Association Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any ECG abnormality at screening has to be documented by the investigator as not medically relevant.
* Pregnant or breastfeeding - methotrexate is Pregnancy Category X - has been reported to cause fetal death and/or congenital abnormalities. Confirmation that the subject is not pregnant must be established by a negative serum beta-human chorionic gonadotropin (beta-hCG) pregnancy test result obtained during screening. Pregnancy testing is not required for post-menopausal or surgically sterilized women.
* Uncontrolled diabetes mellitus defined as a Hemoglobin A1C≥ 10% in patients with a prior history of diabetes, prior to study enrollment.
* Serious concomitant systemic disorders (e.g., active uncontrolled infection or uncontrolled diabetes) or psychiatric disorders that, in the opinion of the investigator, would compromise the safety of the patient or compromise the patient's ability to complete the study.
* Other severe acute or chronic medical or psychiatric conditions, or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for enrollment in this study.
* Any history of epilepsy or a seizure disorder or any known prior seizures.
* Abnormalities on 12-lead electrocardiogram (ECG) considered by the investigator to be clinical significant.
* Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to IGF or methotrexate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2018-02-21 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mrinal S Patniak, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic, Rochester, Minnesota
  - Regions Cancer Care Center, Saint Paul, Minnesota

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | IGF/MTX
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | IGF/MTX
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events
Description: Number of Participants with Treatment-Emergent Adverse Events through study completion, up to a maximum duration of 10 28-day cycles.
Time Frame: Up to 6 28-day cycles for one participant, and up to 10 28-day cycles for the other participant.
Measure: Count of Participants; unit: Participants
Arm/Group | IGF/MTX
Number analyzed (Participants) | 2
Participants | 2

2. Secondary Outcome: Response Criteria for AML, Complete Remission (CR)
Description: Bone marrow blasts, platelet count, independence of red cell transfusions. Bone marrow blasts <5%, absence of blasts with Auer rods, absence of extramedullyary disease, absolute neutrophil count >1.0 x 10(9)/L, independence of red cell transfusions.
Time Frame: Assessed after 2 cycles of 28 days each.
Population: One of the two patients had oligoblastic AML in addition to MDS. Only that one patient is included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | IGF/MTX
Number analyzed (Participants) | 1
Participants | 0

3. Secondary Outcome: Response Criteria for AML, CR With Incomplete Recovery
Description: All CR criteria except for residual neutropenia (<10(9)/L) or thrombocytopenia (<100x 10(9)/L).
Time Frame: Assessed after 2 cycles of 28 days each.
Population: One of the two patients had Oligoblastic AML in addition to MDS. Only that patient is included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | IGF/MTX
Number analyzed (Participants) | 1
Participants | 1

4. Secondary Outcome: Response Criteria for AML, Relapse.
Description: Bone marrow blasts greater the 5% or reappearance of blasts in the blood, or development of extramedullary disease after complete remission or complete remission with incomplete recovery..
Time Frame: Assessed after 6 cycles of 28 days each.
Population: The one patient analyzed achieved complete remission after 2 cycles and relapse after 6 cycles.
Measure: Count of Participants; unit: Participants
Arm/Group | IGF/MTX
Number analyzed (Participants) | 1
Participants | 1

5. Secondary Outcome: Response Criteria for MDS, Complete Remission (CR)
Description: Bone marrow less than 5% myeloblasts with normal maturation of all cell lines. Persistent dysplasia will be noted. Peripheral blood values of Hgb greater than or equal to 11 d/dL, platelets greater than or equal to 100*10^9 platelets/L, neutrophils greater than or equal to 1.0*10^9 neutrophils/L, blasts equal to 0%.
Time Frame: Assessed after 6 cycles of 28 days each.
Measure: Count of Participants; unit: Participants
Arm/Group | IGF/MTX
Number analyzed (Participants) | 2
Participants | 0

6. Secondary Outcome: Response Criteria for MDS, Marrow CR
Description: Bone marrow less than or equal to 5% myeloblasts and decreased by greater than 50% over pretreatment.
Time Frame: Assessed after 2 cycles of 28 days each.
Measure: Count of Participants; unit: Participants
Arm/Group | IGF/MTX
Number analyzed (Participants) | 2
Participants | 1

7. Secondary Outcome: Response Criteria for MDS, Stable Disease
Description: Failure to achieve at least PR, but no evidence of progression for greater than 8 weeks
Time Frame: Assessed after 6 cycles of 28 days each. Both patients had at least stable disease for at least 6 cycles.
Measure: Count of Participants; unit: Participants
Arm/Group | IGF/MTX
Number analyzed (Participants) | 2
Participants | 2

8. Secondary Outcome: Response Criteria for MDS, Failure
Description: Death during treatment or disease progression characterized by worsening of cytopenias, increase in percentage of bone marrow blasts, or progression to a more advanced MDS FAB subtype than pretreatment
Time Frame: Assessed after 6 cycles of 28 days each.
Population: Neither patient met the criteria of failure at any time point (after 2, 4, and 6 cycles of 28 days each).
Measure: Count of Participants; unit: Participants
Arm/Group | IGF/MTX
Number analyzed (Participants) | 2
Participants | 0

9. Secondary Outcome: Response Criteria for MDS, Disease Progression, Blasts Measurements
Description: Absolute blast count.
Time Frame: Assessed after 2 cycles of 28 days each.
Population: 2 subjects overall are analyzed, one subject is analyzed per row of data.
Measure: Number; unit: percentage of bone marrow blasts
Arm/Group | IGF/MTX
Number analyzed (Participants) | 2
percentage of bone marrow blasts
  Subject 101 baseline, 1 participant per row: number analyzed (Participants) | 1
  Subject 101 baseline, 1 participant per row | 22
  Subject 101, 8 weeks, 1 participant per row: number analyzed (Participants) | 1
  Subject 101, 8 weeks, 1 participant per row | 5
  Subject 102 baseline, 1 participant per row: number analyzed (Participants) | 1
  Subject 102 baseline, 1 participant per row | 17
  Subject 102, 8 weeks, 1 partipant per row: number analyzed (Participants) | 1
  Subject 102, 8 weeks, 1 partipant per row | 17

10. Secondary Outcome: Response Criteria for MDS, Disease Progression, Hgb
Description: Hemoglobin in g/dL
Time Frame: Assessed after 2 cycles of 28 days each.
Population: 2 subjects are analyzed overall, but one subject is analyzed per row of data.
Measure: Number; unit: g/dl
Arm/Group | IGF/MTX
Number analyzed (Participants) | 2
g/dl
  Subject 101, baseline, 1 participant per row: number analyzed (Participants) | 1
  Subject 101, baseline, 1 participant per row | 7.3
  Subject 101, 8 weeks, 1 participant per row: number analyzed (Participants) | 1
  Subject 101, 8 weeks, 1 participant per row | 8.9
  Subject 102, baseline, 1 participant per row: number analyzed (Participants) | 1
  Subject 102, baseline, 1 participant per row | 9.7
  Subject 102, 8 weeks, 1 participant per row: number analyzed (Participants) | 1
  Subject 102, 8 weeks, 1 participant per row | 9.9

11. Secondary Outcome: Response Criteria for MDS, Disease Progression, Neutrophils
Description: Neutrophil count in 10(9)/L
Time Frame: Assessed after 2 cycles of 28 days each.
Population: 2 subjects are analyzed overall, but one subject is analyzed per row of data.
Measure: Number; unit: neutrophils x10(9) per liter
Arm/Group | IGF/MTX
Number analyzed (Participants) | 2
neutrophils x10(9) per liter
  Subject 101, baseline, 1 participant per row: number analyzed (Participants) | 1
  Subject 101, baseline, 1 participant per row | 0.04
  Subject 101, 8 weeks, 1 participant per row: number analyzed (Participants) | 1
  Subject 101, 8 weeks, 1 participant per row | 0.75
  Subject 102, baseline, 1 participant per row: number analyzed (Participants) | 1
  Subject 102, baseline, 1 participant per row | 0.38
  Subject 102, 8 weeks, 1 participant per row: number analyzed (Participants) | 1
  Subject 102, 8 weeks, 1 participant per row | 1.29

12. Secondary Outcome: Response Criteria for MDS, Survival, Death
Description: Survival over the full study time period and follow up to 23 months after initiating treatment.
Time Frame: All-cause mortality was assessed up to 23 months, and serious and Other (Not Including Serious) Adverse Events were assessed for up to 22 months.
Population: Number of participants who survived for 23 months.
Measure: Count of Participants; unit: Participants
Arm/Group | IGF/MTX
Number analyzed (Participants) | 2
Participants | 2

ADVERSE EVENTS:
Time Frame: All-cause mortality was assessed up to 23 months, and serious and Other (Not Including Serious) Adverse Events were assessed for up to 22 months.
Arm/Group | IGF/MTX
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 2/2
Other Adverse Events (participants affected / at risk) | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IGF/MTX (N=2)
Subcutaneous abscess (Skin and subcutaneous tissue disorders) | 1 (1) — Subcutaneous abscess from an infection. The adverse event was unrelated to the study medication.
Syncope (Nervous system disorders) | 1 (1) — The syncope was judged possibly study medication related.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IGF/MTX (N=2)
Lymphocyte count decreased (Blood and lymphatic system disorders) | 1 (1) — Grade 3 event. Judged as possibly study medication related.
Worsening anemia (Blood and lymphatic system disorders) | 1 (1) — Grade 3. Judged as possibly study medication related.
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) — Grade 2. Judged as possibly study medication related.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-06): https://cdn.clinicaltrials.gov/large-docs/78/NCT03175978/Prot_SAP_000.pdf